CLINICAL TRIAL: NCT06576518
Title: Exercise Intervention in Patients With Metabolic Syndrome and Renal Disease: a Prospective Study (EXRED)
Brief Title: Exercise Intervention in Patients With Metabolic Syndrome and Renal Disease: a Prospective Study
Acronym: EXRED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of La Laguna (Other)
Collaborators: Fundacion Canaria Instituto de Investigacion Sanitaria de Canarias (Other)
Responsible Party: Principal Investigator, Raúl Morales Febles, PhD-Physiotherapist, University of La Laguna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUC_2021_32
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Metabolic Syndrome; CKD
Keywords: Adherence; Chronic Kidney Disease; Metabolic Syndrome; Obesity; Therapeutic Exercise
MeSH Terms: conditions — Metabolic Syndrome; Renal Insufficiency, Chronic; Obesity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise group (Experimental): Patients with established CKD (1-4) and MS were treated with individualised incremental exercise (aerobic and resistance) for 6 months.
  Interventions: Other: Therapeutic exercise

INTERVENTIONS:
Other: Therapeutic exercise — An individualised incremental exercise programme was simultaneously supported by an adherence plan to assess and promote compliance.

SUMMARY:
INTRODUCTION: Obesity (OB) and metabolic syndrome (MetS) are risk and progression factors for chronic kidney disease (CKD). However, the effect of OB/MetS intervention with exercise on renal function progression and proteinuria is unknown.

OBJECTIVE: To analyse the effect of therapeutic exercise on MetS and main renal outcomes in patients with CKD.

METHODOLOGY: This is a 6-month prospective exploratory study. Patients with stablished CKD (1-4) and MetS were treated with individualised incremental exercise (aerobic and resistance). Simultaneously, a plan of adherence was set up to promote compliance. Renal and metabolic outcomes were collected. The main renal parameters were: proteinuria, in isolated urine samples, and glomerular filtration rate (GFR), measured by iohexol DBS, at 0, 3 and 6 months. At the same time points, metabolic outcomes were measured: weight, dyslipidemia, insulin resistance and hypertension.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* CKD of diverse aetiologies
* estimated GFR ≥ 30 ml/min
* BMI ≥ 27 kg/m2 associated to MetS or diabetes mellitus (DM)
* stable renal function for at least 6 months before screening
* ability to perform exercise

Exclusion Criteria:

* clinical conditions that exclude exercise therapy such as clinical instability, active infection, cancer, acute cardiovascular disease, advanced CKD, pulmonary hypertension, or limb amputations
* inability to understand the protocol
* severe psychiatric illness
* allergy to iodine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Changes in Glomerular filtration rate (GFR) and urine abulmin-creatinine ratio (UACR). | Baseline, 3 and 6 months
  GFR and UACR were measured at baseline, 3 and 6 months, with the gold standard method of plasma clearance of iohexol (DBS technique) and urine analysis (isolated urine samples), respectively. The researchers expect a change in terms of GFR (improvement of hyperfiltration) and UACR reduction compared to baseline.

SECONDARY OUTCOMES:
Changes in body weight and MetS traits (Analytics). | Baseline, month 3 and 6.
  Monthly, weight in kilograms, height in meters, waist circumference, hip circumference, will be measured. Also, BMI Body mass index (BMI): weight in kilograms divided by the square of the height in meters.Weight changes >5% were expected at 6 months.
  Changes in Mets traits as a relative change from baseline (%) or as success in falling below the cut-off point of the MetS definition. To evaluate the improvements in metabolic risk factors profile: obesity, triglycerides, blood pressure and HDL cholesterol.hemogram (hematocrit, haemoglobin, white blood count), biochemist tests: creatinine, HbA1c, total, LDL and HDL cholesterol, triglycerides, uric acid, hepatic enzymes (ASAT, ALAT), levels of immunosuppression, albumin, creatinine, albuminuria, proteinuria in an isolated urinary samples.
Compliance-adherence | Monthly
  To ensure compliance, the following measures will be implemented: (a) contact by phone one time per week, (b) individual interview every month to reinforce lifestyle changes and follow all recommended in the exercise prescription; (c) the use of a gadget (xiaomi mi band) to see daily routines of patients and every training prescription, analysing the time, frequency, burned calories, velocity and distance, among others, to reach the established goal prescribed by the physiotherapist.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de La Laguna, San Cristóbal de La Laguna, Santa Cruz De Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rivero Martin O, Morales Febles R, Delgado Mallen PI, Reseghetti E, Miquel Rodriguez RM, Estupinan Torres S, Cobo Caso MA, Cruz C, Diaz Martin L, Gonzalez Martin AR, Sanchez Baez DJ, Hernandez Marrero DJ, Luis Lima S, Porrini E. Exercise Intervention in Patients with Metabolic Syndrome and Renal Disease: A Prospective Study (EXRED). Nephron. 2025 Nov 27:1-15. doi: 10.1159/000549072. Online ahead of print. PMID 41308049